CLINICAL TRIAL: NCT03041480
Title: The Association Between Periodontal Status, Serum Lipid Levels and Lipoprotein Associated Lipophosphase A2(Lp-PLA2) in Chronic Periodontitis Subjects and Healthy Controls: A Case Control Study
Brief Title: Serum Lipid Levels and Lp-PLA2 in Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB/2015/91
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Periodontitis (Disorder)
Keywords: chronic periodontitis; lipids; Lp-PLA2
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GROUP I: Estimation of serum lipid levels and Lp-PLA2 in generalized severe chronic periodontitis
  Interventions: Diagnostic Test: serum lipid levels and Lp-PLA2
- GROUP II: Estimation of serum lipid levels and Lp-PLA2 in generalized moderate chronic periodontitis
  Interventions: Diagnostic Test: serum lipid levels and Lp-PLA2
- GROUP III: Estimation of serum lipid levels and Lp-PLA2 in systemically and periodontally healthy controls
  Interventions: Diagnostic Test: serum lipid levels and Lp-PLA2

INTERVENTIONS:
Diagnostic Test: serum lipid levels and Lp-PLA2 — Estimation of Total Cholesterol, triglyceride, High density lipoprotein, Low density lipoprotein, very low density lipoprotein and Lipoprotein associated lipophosphase A2 in chronic periodontitis
  Other Names: Biological marker

SUMMARY:
To assess the association between periodontal parameters, serum lipid profile and Lp-PLA2 level in systemically healthy Chronic Periodontitis subjects and healthy controls.

DETAILED DESCRIPTION:
Seventy five participants were divided into 3 groups. The groups consisted of GROUP I- generalized severe chronic periodontitis, GROUP II- generalized moderate chronic periodontitis and GROUP III- systemically and periodontally healthy volunteers who served as control. The selected patients were then evaluated for periodontal parameters, lipid profile and Lp-PLA2.

ELIGIBILITY:
Inclusion Criteria:

Group I:

1. Subjects with age ≥ 35 years.
2. Presence of at least 24 teeth, with Clinical attachment loss (CAL) ≥ 5mm in more than 30% of sites.

Group II:

1. Subjects with age ≥ 35 years.
2. Presence of at least 24 teeth, with Clinical attachment loss (CAL) between 3-4 mm in more than 30% of sites.

Group III:

1. Subjects with age ≥ 35 years.
2. Healthy and intact periodontium

Exclusion Criteria:

1. Presence of any systemic disease or conditions that could affect periodontal tissues.
2. History of periodontal treatment in past 6 months.
3. Smoking and alcoholism
4. Anomalies of blood and immune system
5. Systemic medication or antibiotic treatment for the previous 6 months.
6. Pregnant females.

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population was selected from the Department of Periodontology, Meenakshi Ammal Dental College
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2015-08-23 (Actual); Study Completion 2015-11-26 (Actual)

PRIMARY OUTCOMES:
Estimation of serum Lp-PLA2 | 9 months
  Serum Lp-PLA2 was estimated in all the groups using ELISA

SECONDARY OUTCOMES:
Estimation of serum lipid profile | 9 months
  Serum Total cholesterol, triglyceride, High density lipoprotein, Low density lipoprotein and very low density lipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Bittu Koshy, BDS, Principal Investigator — Meenakshi Ammal Dental College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou SY, Xiao WM, Ouyang XY. Lipoprotein-associated phospholipase A2 and serum lipid levels in subjects with chronic periodontitis and hyperlipidemia. Chin J Dent Res. 2012;15(1):25-9. PMID 22866279
- [Background] Fentoglu O, Koroglu BK, Kara Y, Dogan B, Yilmaz G, Sutcu R, Ay ZY, Tonguc MO, Orhan H, Tamer MN, Kirzioglu FY. Serum lipoprotein-associated phospholipase A(2) and C-reactive protein levels in association with periodontal disease and hyperlipidemia. J Periodontol. 2011 Mar;82(3):350-9. doi: 10.1902/jop.2010.100417. Epub 2010 Sep 1. PMID 20809860